CLINICAL TRIAL: NCT00006148
Title: Spleen Size in Peripheral Blood Stem Cell Donors
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000192; 00-CC-0192
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-06

CONDITIONS: Splenomegaly
Keywords: Granulocyte Colony - Stimulation Factor; Peripheral Blood Stem Cells; Splenomegaly
MeSH Terms: conditions — Splenomegaly

SUMMARY:
This study will determine whether the spleen in people who donate stem cells (bone marrow cells collected from the blood) enlarges as a result of taking granulocyte colony-stimulating factor (G-CSF). Donors take this growth factor to maximize the amount of stem cells that can be collected for transplantation to patients with leukemia or other diseases. The study will also examine whether changes in the donor's white blood cell count, blood stem cell count, and blood chemistries can predict a change in spleen size.

Stem cells donors take G-CSF for 5 to 6 days before donating. Besides increasing the number of stem cells and white blood cells in the bloodstream, the drug also causes some other temporary changes in blood chemistry. Many people who take G-CSF for a few days get a headache, feel an ache in their bones, or feel tired for a few days. About one-third of patients chronically treated with G-CSF to raise blood cell counts develop an enlarged spleen. It is not known if a brief 5- to 6-day course of G-CSF also affects the size of the spleen, but about 1 in 10,000 blood stem cell donors have had a spontaneous rupture of the spleen.

Adults and children 18 years of age and older who are donating stem cells for relatives enrolled in clinical trials at the National Institutes of Health may participate in this study. They will donate stem cells according to the standard procedure, but will give an extra 15 milliliters (3 teaspoons) of blood both before receiving G-CSF and after donating stem cells. Donors' spleen size will be measured by ultrasound scanning of the abdomen three times: the day before receiving G-CSF, the day after donating the stem cells and 4 days after donating.

DETAILED DESCRIPTION:
The administration of granulocyte-colony stimulating factor (G-CSF) leads to splenic enlargement in approximately one third of neutropenic patients who are chronically treated with this drug. Short courses, 5 to 6-days, of G-CSF are used to increase the yield of hematopoietic progenitor cells collected by apheresis from peripheral blood stem cell (PBSC) donors. G-CSF mobilized PBSC concentrates are increasingly replacing marrow as a source of hematopoietic progenitor cells for transplants involving HLA-compatible relatives. PBSC donors experience splenomegaly and rarely, spontaneous rupture of the spleen. Since splenomegaly is a risk factor for splenic rupture, it is important to determine the incidence and time course of splenic enlargement in PBSC concentrate donors. This protocol will prospectively study 40 subjects donating G-CSF mobilized PBSC for HLA compatible relatives or donating PBSC's for laboratory investigations at the Department of Transfusion Medicine in the Warren G. Magnuson Clinical Center. The subjects will be given G-CSF for 5 days and a PBSC concentrate will be collected on day 5. Ultrasound scans will be used to assess their spleen size. The scans will be performed before G-CSF administration and the day the last PBSC concentrate is collected. A third scan will be performed 10 or 11 days after the last PBSC is collected. The effects of several parameters on spleen size will be assessed including: donor age, gender, race and changes in liver function assays, white blood cell counts, platelet counts, and CD34+ cell counts.

ELIGIBILITY:
INCLUSION CRITERIA

Adults and children 18 years of age or greater will be studied.

Enrolled in a primary stem cell transplant protocol that has been approved by the IRB.

Potential subjects are people donating PBSC concentrates for HLA-compatible relatives as part of IRB approved protocols or donating PBSCs for laboratory investigations.

EXCLUSION CRITERIA

Donors who cannot remain in the Bethesda area for an additional 4 to 5 days following their donations will be excluded from the third ultrasound.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49
Dates: Start 2000-08; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bensinger WI, Weaver CH, Appelbaum FR, Rowley S, Demirer T, Sanders J, Storb R, Buckner CD. Transplantation of allogeneic peripheral blood stem cells mobilized by recombinant human granulocyte colony-stimulating factor. Blood. 1995 Mar 15;85(6):1655-8. PMID 7534140
- [Background] Korbling M, Przepiorka D, Huh YO, Engel H, van Besien K, Giralt S, Andersson B, Kleine HD, Seong D, Deisseroth AB, et al. Allogeneic blood stem cell transplantation for refractory leukemia and lymphoma: potential advantage of blood over marrow allografts. Blood. 1995 Mar 15;85(6):1659-65. PMID 7888684
- [Background] Schmitz N, Dreger P, Suttorp M, Rohwedder EB, Haferlach T, Loffler H, Hunter A, Russell NH. Primary transplantation of allogeneic peripheral blood progenitor cells mobilized by filgrastim (granulocyte colony-stimulating factor). Blood. 1995 Mar 15;85(6):1666-72. PMID 7534141